CLINICAL TRIAL: NCT04438954
Title: Investigation of Fatigue, Physical Activity, Sleep Quality and Anxiety Levels of Multiple Sclerosis Patients in the COVID-19 Pandemic
Brief Title: Investigation of Fatigue, Physical Activity, Sleep Quality and Anxiety Levels
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis; Covid-19
Keywords: Multiple Sclerosis; Covid-19 pandemic; Fatigue; Physical activity; Sleep quality; Anxiety
MeSH Terms: conditions — Multiple Sclerosis; COVID-19; Fatigue; Motor Activity; Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hundreds of thousands of confirmed cases have been reported worldwide, just 3 months after the first patients were identified in Wuhan, China. Just like other members of the community, MS patients are uncomfortable with the emotional distress and health anxiety caused by the COVID-19 outbreak. Most MS patients receive immunosuppressive or immunomodulatory therapies. Patients taking immunosuppressive agents are theoretically at increased risk of being affected by viral pandemics, and a higher health concern is expected in this group of patients. Moreover, MS patients lose social support. Patients with increased duration of stay can no longer access physical and cognitive rehabilitation therapies. We also know that increased anxiety and sleep disorders can cause MS patients to have an attack.

When literature is examined, it is known that MS patients' physical activity levels decrease, fatigue, sleep quality and anxiety levels increase, so their quality of life and participation in daily life activities decrease. MS patients lose social support during the COVID-19 outbreak. For all these reasons, we think that the fatigue, physical activity level, anxiety level and sleep disturbances affected before the COVID-19 outbreak will be further affected for these reasons.

ELIGIBILITY:
Inclusion Criteria:

* patients with a confirmed diagnosis of clinically definite MS, physician-administered Expanded Disability Status Scale (EDSS) range of 1-5, and following the instructions.

Exclusion Criteria:

* patients with acute attacks (three months prior to the study) and those included on the physiotherapy program during the Covid-19 pandemic.

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Fatigue | 4 week
  Fatigue was assessed by the Fatigue Severity Scale (FSS). This is a 9-item questionnaire that assesses the effect of fatigue on daily living. Each item is a statement on fatigue that the subject rates from 1 "completely disagree" to 7 "completely agree". A score of 4 or higher generally indicates severe fatigue
Physical activity | 4 week
  Physical activity levels were assessed by the International Physical Activity Questionnaire (IPAQ): short form. The online self-reporting questionnaire consisted of questions investigating the respondents' PA practice in terms of frequencies and durations of sitting, walking, moderate-intensity physical activities and vigorous-intensity physical activities. The MET-minutes per week (MET-min/week) were calculated using the following formula: intensity (MET) x duration x frequency. Physical activity levels were classified as physically inactive (<600 MET-min/week), with low levels of physical activity (600-3000 MET- min/week) and physical activity level that is sufficient (> 3000 MET-min/week)
Sleep quality | 4 week
  The Pittsburgh Sleep Quality Index (PSQI) questionnaire was used to measure sleep quality using an 18-item scale containing seven items that included sleep quality, sleep duration, sleep latency, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction. Each dimension scored between 0-3, with a total score ranging from 0-21, and a higher score indicating lower sleep quality.
Anxiety | 4 week
  The Hospital Anxiety and Depression Scale (HADS) was composed by two subscales (i.e., anxiety and depression), with 7-items each. The anxiety part of HADS was used to evaluate the anxiety levels of the patients. Each dimension scored between 0-3, with a total score ranging from 0-21, and a higher score indicating higher anxiety level.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)